CLINICAL TRIAL: NCT01025219
Title: A Case Control Study on Contribution to the Analysis of the Phenotypic Heterogeneity in Crack/Cocaine Addiction
Brief Title: A Contribution to the Analysis of the Phenotypic Heterogeneity in Crack/Cocaine Addiction : a Case Control Study
Acronym: CRACK-ANT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Center of Martinique (Other)
Responsible Party: RIAM Daniel, CHU de Fort-de-France
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 09/B/01
Record Dates: First submitted 2009-12-01; First posted 2009-12-03 (Estimated); Last update posted 2011-03-22 (Estimated); Status verified 2011-03

CONDITIONS: Dependence, Cocaine
Keywords: Diagnosis of dependence on cocaine according to DSM-IV-TR criteria
MeSH Terms: conditions — Cocaine-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Genetic: Collect 10 ml of Saliva for DNA extraction — After signed written informed consent, all patients and controls have clinical and neuropsychological evaluations (DIGS, WURS, BROWN, BIS, SSS and IGT) for phenotypic diagnosis and collection of saliva for DNA extraction and genotyping diagnosis.

SUMMARY:
The purpose of this study is to assess the phenotypic candidates symptoms, in patients with crack/cocaine addiction, in terms of clinical comorbidities, dimensions of personality, and neuropsychological evaluations apt to be associated with genetic and genotypic characterisations, notably on the polymorphisms of the genes coding or regulating dopaminergic, norepinephrine and serotoninergic systems.

DETAILED DESCRIPTION:
Genetic studies show an association between drug addiction and the dopaminergic system and its modulators. Nonetheless, results are contradictory, partially due to the heterogeneity of the phenotype addiction. Placed on the trafficking route of cocaine, and homogeneously populated, Martinique is of particular interest for the study of the vulnerability of the crack/cocaine addiction. In a precedent study, supported by a grant MILDT / INSERM 2000, on 155 men dependent to crack/cocaine and characterised with three clinical dimensions -sensation seeking, impulsivity and childhood ADHD- we found an association between each dimension and polymorphisms of DRD2 and DRD4 genes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cocaine abuse/dependence according to DSM-IV-TR criteria
* Come from French West Indies (3 grandparents are African-Caribbean)
* Sign a written informed consent

Exclusion Criteria:

* Minor
* Men with no cocaine abuse/dependence according to DSM-IV-TR criteria

For the control:

Inclusion Criteria:

* Platelets donor
* No substance abuse/dependence according to DSM-IV-TR criteria
* Come from French West Indies (3 grandparents are African-Caribbean)
* Sign a written informed consent

Exclusion Criteria:

* Minor
* Men refusing a genetic study

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2009-12; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The specific measure that will be related to core objectives of the study is to constitute a sample collection from saliva. | The saliva will be collect at the end of the first visit

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme LACOSTE, MD, Principal Investigator — CHU de Fort-de-France
Locations (1):
- Service de psychiatrie et addictologie - CHU de Fort-de-France, Fort-de-France, Martinique, France